CLINICAL TRIAL: NCT06177847
Title: Efficacy of BIS Monitoring in Deep Hypnotic State and Its Outcome on Patient Undergoing Elective Neurosurgery
Brief Title: Efficacy of BIS Monitoring in Deep Hypnotic State
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Bintang Pramodana, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaU432
Record Dates: First submitted 2023-09-21; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Hypnotic; Withdrawal State With Delirium; Neurological Disorder; Postoperative Delirium; Postoperative Confusion; Anesthesia; Anesthesia Emergence Delirium; Gas; Inhalation
Keywords: Deep Hypnotic State; Anesthesia; Postoperative complication; Neurosurgical disorder
MeSH Terms: conditions — Nervous System Diseases; Emergence Delirium; Mucopolysaccharidosis IV; Respiratory Aspiration; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: In the group with BIS where the anesthesia protocol is opened, namely the use of anesthetic gas, the anesthetic drug will be adjusted to the BIS value range of 40-60 or BIS-guided
Who Masked: Participant, Care Provider
Masking Description: The anesthesia protocol used in closed BIS is carried out like general anesthesia without using BIS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BIS Guided (Experimental): In the group with BIS where the anesthesia protocol is opened, namely the use of anesthetic gas, the anesthetic drug will be adjusted to the BIS value range of 40-60 or BIS-guided
  Interventions: Device: BIS
- BIS Blinded (No Intervention): The anesthesia protocol used in closed BIS is carried out like general anesthesia without using BIS.

INTERVENTIONS:
Device: BIS — In the group with BIS where the anesthesia protocol is opened, namely the use of anesthetic gas, the anesthetic drug will be adjusted to the BIS value range of 40-60 or BIS-guided
  Arms: BIS Guided

SUMMARY:
Determining the efficacy of the BIS monitor in monitoring deep hypnotic states as well as intra- and post-operative outcomes in neurosurgery patients

DETAILED DESCRIPTION:
This study will be conducted with a two-group, double-blind, randomized clinical trial design in elective patients who will undergo neurosurgical procedures under general anesthesia. Patients scheduled for elective neurosurgery who meet the inclusion criteria will be randomized into one of the intervention groups, with or without BIS. Demographic data will be taken from medical records. In both groups, the BIS probe will be inserted before induction, but for the control group, the BIS monitor will be closed, while for the intervention group, anesthesia will be titrated according to the BIS value to maintain the BIS value in the range of 40-60. In the group with an open BIS, the anesthesia protocol is the use of anesthetic gas, and the anesthetic drug will be adjusted to the BIS value range of 40-60 or BIS-guided, while the anesthesia protocol used in a closed BIS is carried out like general anesthesia without using BIS. The BIS value will be recorded minute by minute according to the extraction feature of the BIS machine after surgery. The total use of anesthetic agents, duration of surgery, and intraoperative hemodynamics will be recorded through anesthesia status. The patient will follow the progress until the patient is discharged from the hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-60 years with an ASA tolerance of 1-2 who will undergo general anesthesia techniques
* Operation duration > 3 hours
* The patient agrees to take part in the study.

Exclusion Criteria:

* Continuous intraoperative use of ketamine, magnesium sulfate, dexmedetomidine, lidocaine agents
* Massive bleeding that causes hemodynamic disturbances
* Severe electrolyte disturbances
* Severe liver or kidney function disorders
* The patient was decided not to extubate in the operating room

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Deep Hypnotic State | During surgery and up to 24 hours after surgery
  the state of depth of anesthesia where the Bispectral Index value is <40. is calculated from the beginning of induction to the end of the operation and accumulated at the end of the operation.
Total use of anesthetic agents | During surgery and up to 24 hours after surgery
  The amount of anesthetic gas used from the start of the operation to the end of the operation
Number of Participants with Hypotension and Bradycardia Intraoperative | During surgery and up to 24 hours after surgery
  Intraoperative hypotension was defined as systolic blood pressure <90 mm Hg for >5 minutes or a 35% decrease in MAP. Intraoperative bradycardia was defined as a heart rate <60 beats/min for >5 minutes
Vasopressor use | Before surgery, during surgery, up to 24 hours after surgery
  Use of vasopressor agents (dopamine, dobutamine, norepinephrine, epinephrine, etc.) will be calculated and totaled at the end of surgery.
Incidence of delirium | up to 24 hour after surgery
  The method for measuring the incidence of delirium will be assessed by researchers using the CAM (Confusion Assessment Method) questionnaire which has been validated in Indonesian
Incidence of mortality | up to 28 days after surgery
  The incidence of death after surgery in hospital or outside the hospital
Lenght of stay | From the date of randomization until 28 days after surgery
  The length of stay is measured from days after surgery until being discharged from the hospital.
Duration of recovery | up to 7 days post operative
  The duration of recovery was measured from post-operative day 0 until the patient was able to return to the patient's baseline function